CLINICAL TRIAL: NCT04468204
Title: Use of Novel Sinusonic Device for Prevention of Community Acquired Upper Respiratory (URI)
Brief Title: Use of Novel Sinusonic Device for Prevention of Community Acquired Upper Respiratory Infection (URI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Shaun A. Nguyen, MD, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00100980
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Upper Respiratory Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SinuSonic Device (Experimental): SinuSonic device used for 1 min three times a day for 8 weeks.
  Interventions: Device: SinuSonic Device
- Sham (Sham Comparator): Sham SinuSonic device used for 1 min three times a day for 8 weeks.
  Interventions: Device: Sham SinuSonic Device

INTERVENTIONS:
Device: SinuSonic Device — A medical device that utilizes sound and pressure combined with normal breathing to relieve nasal congestion.
  Arms: SinuSonic Device
Device: Sham SinuSonic Device — Sham positive expiratory pressure intervention using the SinuSonic Device.
  Other Names: Sham
  Arms: Sham

SUMMARY:
This study aims to test the safety, efficacy and potential mechanism of action of the SinuSonic device on adults with upper respiratory infection (URI). SinuSonic is a medical device that utilizes sound and pressure combined with normal breathing. The study will have 2 aims. Aim 1 willdetermine if Sinusonic decreases the number of URIs experienced during an 8 week fall URI season. Subjects will use an active device (positive expiratory pressure and 128 Hz) or a sham device (no positive expiratory pressure and 1,000 Hz) for 1 min tid for 8 weeks. Aim 2 will determine if Sinusonic decreases the severity and duration of community acquired viral URIs. Subjects will use active or sham device as above.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older with no transient symptoms of any URI or allergies at baseline.

Exclusion Criteria:

* Any transient ENT condition that may impact upper airway to include acute sinusitis or otitis.
* Any upper respiratory illness within last 2 weeks
* TSS will be measured at baseline as described above and must be <9 for inclusion (Eccles etal).
* Topical decongestant use in last week
* Current nasal crusting or history of ulceration or perforation
* History of severe nose bleeding within last 3 months
* Known pregnancy
* Immunosuppressed condition or on immune modulating medications such as prednisone or chemotherapy
* Allergic sensitivity to silicone or any other component of device
* Inability to read and understand English
* Inability to perform treatment due to underlying medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sinus Center - Medical Univesity of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Not Applicable. The investigators plan to publish this study.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SinuSonic Device | Sham
Started | 39 | 13
Completed | 39 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SinuSonic Device | Sham | Total
Number analyzed (Participants) | 39 | 13 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 12 | 47
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Full Range); unit: years] | 46.2 [20 to 69] | 48.5 [39 to 69] | 46.8 [20 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 7 | 34
  Male | 12 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 38 | 13 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 39 | 11 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Symptoms Score (TSS)
Description: The Total Symptom Score (TSS) was based on the severity of each of upper respiratory infection (URI) symptom.
  The TSS includes 9 symptoms: Lost sense of smell/taste, sneezing, runny nose or thick nasal discharge, nasal obstruction or congestion, sore throat, cough headache, maliase, and chilliness.
  The severity of URI symptoms was scored on a symptom severity scale (0 = not at all; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms)
  Minimum score=0; maximum score=27.
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | SinuSonic Device | Sham
Number analyzed (Participants) | 39 | 13
scores | 0.503 (0.501) | 0.843 (0.569)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | SinuSonic Device | Sham
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/13
Other Adverse Events (participants affected / at risk) | 1/39 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SinuSonic Device (N=39) | Sham (N=13)
Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT04468204/Prot_SAP_000.pdf